CLINICAL TRIAL: NCT01537848
Title: Retrospective Study of Endoscopic Ultrasound Guided Transmural Drainage of Post-operative Collections
Brief Title: Retrospective Study of Endoscopic Ultrasound (EUS) Guided Transmural Drainage of Post-operative Abdominal Collections
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Lemmers Arnaud, MD, PhD, Erasme University Hospital
Other Study IDs: EUS in surgical collection; P2012/059 (Other: Erasme Hospital Ethics Committee)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Post-surgical Intra-abdominal Collection
Keywords: EUS; Endoscopic ultrasound; abdominal collection; post-operative; post-surgical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- post-operative collection: patients suffering from a post-operative abdominal collection
  Interventions: Procedure: EUS guided transmural drainage

INTERVENTIONS:
Procedure: EUS guided transmural drainage — Puncture of the collection is done under EUS guidance using a linear echoendoscope (FG-3830UT, Pentax or Olympus GF-UCT140/180 or forward viewing scope (Olympus)) with a 19G echoTip needle or a cystotome (Cook Medical Inc.). Then a 0.035 guidewire is inserted in the collection and the hole is enlarged with a cystotome (Cook Medical) or a 6.5F diathermic sleeve (Endoflex) and sometimes if needed a 6-8mm CRE balloon (Boston Scientific) before stenting with one or two double pigtail plastic stents (Cook Endoscopy, Endoflex). A nasocystic drain was also put whenever needed. If only a single stent could be placed in the first attempt, a subsequent procedure is scheduled for insertion of additional stents after dilation of the tract. There isn't any specific drug given during the procedure.
  Other Names: Echoendoscope (Pentax FG-3830UT; Olympus GF-UCT140/180); 19G echoTip needle (Cook Medical); Cystotome (Cook Medical); diathermic sleeve (Endoflex); CRE balloon (Boston Scientific); double pigtail stents (Cook Endoscopy, Endoflex)

SUMMARY:
This is a retrospective study of a single center on endoscopic ultrasound (EUS) guided transmural drainage of post-operative collections during a 9 years period.

DETAILED DESCRIPTION:
All patients who underwent a EUS guided drainage of post-operative collection between 2002 and 2011 in the endoscopy unit of Erasme hospital will be included for analysis. The study will focus on retrospective analysis of prospectively collected data. The technique is the same as the one used for pancreatic pseudocysts drainage. The technical success is defined as the ability to access and drain the collection by placement of transmural drain and/or stents. Treatment success (regression of collection) is defined as the resolution of the collection as shown on abdominal imaging (CT or MRI) in association with clinical resolution of symptoms at 8 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent EUS guided drainage of post-operative collections admitted between january 2002 and july 2011 for this treatment in the endoscopic department of a single academic center will be included for analysis.

Exclusion Criteria:

* none (patients for whom other modalities of fluid drainage failed were also included in the study

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent EUS guided drainage of post-operative collections admitted between january 2002 and july 2011 for this treatment in the endoscopic department of a single academic center will be included for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2002-01; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Treatment success | 8 weeks after treatment
  Regression of collection = resolution of collection as shown on abdominal imaging (Ct or MRI) in association with clinical resolution of symptoms at 8 weeks of follow-up

SECONDARY OUTCOMES:
technical success | day of procedure (day 1)
  Success to access and drain the collection by the placement of transmural drain and/or stent(s)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Devière, MD,PhD, Study Chair — Erasme Hospital, ULB (Université Libre de Bruxelles), Belgium
Locations (1):
- Erasme Hospital, Gastroenterology Department, ULB (Université libre de Bruxelles), Brussels, Belgium